CLINICAL TRIAL: NCT05346640
Title: Augmenting Gait in a Population Exhibiting Foot Drop With Adaptive Functional Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cionic, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Webster, Clinical Operations, Cionic, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIONIC-001
Record Dates: First submitted 2022-04-11; First posted 2022-04-26 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Foot Drop
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Intervention Model Description: A one-group, pre-test post-test study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional electrical stimulation in individuals with foot drop (Experimental): Comparison of kinematics in stimulated and unstimulated gait using functional electrical stimulation in individuals with foot drop as a result of a neurological dysfunction
  Interventions: Device: Cionic Neural Sleeve

INTERVENTIONS:
Device: Cionic Neural Sleeve — Adaptive, functional electrical stimulation

SUMMARY:
The objective of this study is to investigate the effects of personalized, adaptive, current-steering functional electrical stimulation (FES) of the lower leg to improve gait in people with foot drop.

DETAILED DESCRIPTION:
Adaptive, current-steering FES enables precise control over dorsiflexor and evertor muscles, allowing for personalized treatment to correct key foot drop characteristics including dorsiflexion at heel strike and ankle inversion during swing phase. All participants will receive adaptive FES of the dorsiflexors and evertors during back-to-back walking sets. Participants completed up to three walking sets of unstimulated walking (pre-test) followed by lower-leg stimulated walking (post-test). The primary outcome measures include ankle dorsiflexion at heel strike and mean ankle inversion during swing phase. Secondary outcome measures include foot angle at heel strike and single-side heel strike to toe strike time (heel-toe time).

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-70

* Lower extremity impairment that makes walking difficult or uncomfortable
* Capable of sitting, standing, and walking independently or with assistance
* Able to walk at least 50 feet independently or with assistance
* Able to understand and follow basic instructions in English

Exclusion Criteria:

* Have non-reversible damage to the peripheral nervous system
* Have underlying pre-existing conditions like thrombosis/hemorrhage, severe epilepsy or other seizure disorder, severe atrophy or history of implanted electrical devices
* Have cognitive impairment that would prevent you from fully understanding the study and ability to provide informed consent
* Have lower motor neuron disease or injury that may impair response to stimulation
* Are pregnant
* Are under the age of 18 years old
* Have skin conditions of the affected lower limb, including cuts, burns or lesions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cionic, Inc., San Francisco, California
  - Cleveland State University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
Started | 60
Completed | 32
Not Completed | 28
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 14
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physiological Complications | 3
Not completed — Other Reason | 3

BASELINE CHARACTERISTICS:
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.1)
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2
  40-49 years | 3
  50-59 years | 10
  60-69 years | 11
  70-79 years | 5
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diagnosis [Count of Participants; unit: Participants]
  Stroke | 20
  Multiple Sclerosis | 8
  Cerebral Palsy | 1
  Spinal Injury | 2
  Idiopathic | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Dorsiflexion at Heel Strike
Description: Dorsiflexion measured via inertial measurement unit (IMU) sensors placed on the foot and lower leg, measured in degrees. Heel strike is determined from pressure sensors in the shoe.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
Number analyzed (Participants) | 32
degrees | 5.2 [3.5 to 6.8]

2. Primary Outcome: Mean Ankle Inversion During Swing Phase
Description: Ankle inversion measured via IMU sensors placed on the foot and lower leg, measured in degrees. Swing phase is determined from pressure sensors in the shoe
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
Number analyzed (Participants) | 32
degrees | -3.6 [-5.3 to -1.8]

3. Secondary Outcome: Mean Foot Angle at Heel Strike
Description: Foot angle measured via IMU sensors placed on the foot and lower leg, measured in degrees. Heel strike is determined from pressure sensors in the shoe.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
Number analyzed (Participants) | 32
degrees | 5.5 [3.9 to 7.0]

4. Secondary Outcome: Mean Heel-Toe Time as a Percent of Gait Cycle
Description: Time of heel-toe, or single-side heel strike to toe strike measured by percent of gait, where 0% represents heel strike and 100% is the next heel strike. Heel strike assessed by pressure sensors placed in the shoe.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: percentage of gait cycle
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
Number analyzed (Participants) | 32
percentage of gait cycle | 3.4 [1.9 to 4.8]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Functional Electrical Stimulation in Individuals With Foot Drop
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
This study did not include the collection of certain traditional gait analysis metrics including spatial measures like gait speed and stride length as we relied solely on the on-body device for all data collection and metric extraction. Additionally, we were not able to compare functional electrical stimulation treatment impacts relative to standard of care, i.e. ankle-foot orthosis, in a randomized control trial (RCT). An RCT remains a future research study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT05346640/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT05346640/SAP_001.pdf